CLINICAL TRIAL: NCT03492138
Title: A Phase I/II Study of the Addition of Ixazomib to ONC201 and Dexamethasone in Relapsed and/or Refractory Multiple Myeloma
Brief Title: Ixazomib, ONC201, and Dexamethasone in Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Ajai Chari (Other)
Responsible Party: Sponsor-Investigator, Ajai Chari, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 17-2680
Record Dates: First submitted 2018-03-22; First posted 2018-04-10 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Relapsed and Refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — TIC10 compound; ixazomib; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Single arm, open-label, standard 3+3 phase 1 with a Simon 2-stage design followed by stage 2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with relapsed/refractory multiple myeloma (Experimental): ONC201, ixazomib, and dexamethasone in relapsed/refractory multiple myeloma. Run-in phase of ONC201 and dexamethasone weekly until progression at 4 weeks, lack of response at 8 weeks, or progression followed by the addition of weekly ixazomib.
  Interventions: Drug: ONC201; Drug: Ixazomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: ONC201 — 625mg
Drug: Ixazomib — Dose to be determined in Phase 1 of study
Drug: Dexamethasone — 40mg

SUMMARY:
ONC201 is a novel dopamine receptor D2 antagonist that is able to activate the integrated stress response pathway. It is active against multiple myeloma cells in vitro, both as a single agent and in combination with corticosteroids and proteasome inhibitors. In order to document superiority over the combination compared to the individual agents of ixazomib and ONC201 in a single arm study, there will initially be a run-in period of weekly ONC201 625 mg with dexamethasone 40 mg such that if there is progression of disease (25% increase) after 4 weeks or less than a minimal response (25% reduction) after 8 weeks then ixazomib will be added. Dexamethasone is dose-reduced to 20 mg at the same schedule for subjects ≥ 75 years old. If patients do achieve single-agent responses with ONC201 (minimal response or better), they will continue with weekly ONC201 and dexamethasone until progression, with response assessments after each 28-day cycle. Patients who have previously been treated on another clinical trial with weekly ONC201 625mg with dexamethasone with progression while receiving treatment do not need to complete the run-in phase of the study.

At the time of progression, they will proceed to the 3 drug combination phase of the study. It is at the point of 3 drug initiation, that below phase I DLT principles or phase II disease control rate considerations apply.

DETAILED DESCRIPTION:
Phase I Study Design

• Phase I will follow a 3+3 dose escalation design to determine the RPTD of ixazomib in combination with ONC201 and Dexamethasone.

The dose escalation rules for the phase I portion of the study are as follows, escalating in cohorts of 3 patients per dose level including a de-escalation option in case of early toxicity. Dose limiting toxicity (DLT) is defined as any grade 3 or higher toxicity seen during the first 28 day cycle of the triplet regimen (ONC201, ixazomib, and dexamethasone). Of note, grade 3 and higher absolute lymphopenia and hematologic toxicities without clinical sequelae (eg. neutropenia without fever/infection, anemia without symptoms, thrombocytopenia without bleeding) and also responsive to growth factors/transfusions will not be considered DLTs. AST or ALT values of ≥ 3x ULN AND with serum total bilirubin level of > 2x ULN or international normalized ratio (INR) > 1.5 without signs of cholestasis and with no other clear alternative reason to explain the observed liver-related laboratory abnormalities is also considered a DLT. Three patients will be treated at the current dose level. If at least 2 patients are observed to have a DLT, the prior dose level is defined as the RPTD unless only 3 patients have been treated at that level, in which case it is the tentative RPTD. If 0 of the 3 patients are observed to have DLT, the dose level is escalated one dose level for the next cohort of 3 patients, and the process continues as above. If exactly 1 of the 3 patients treated show DLT, 3 additional patients are treated at the current dose level. If none of these additional 3 patients show DLT, the dose level is escalated for the next cohort of 3 patients, and the process continues as above; otherwise, the prior dose level is defined as the RPTD (unless only 3 patients have been treated at that level, in which case it is the tentative RPTD). A tentative RPTD becomes final when a total of 6 patients are treated with less than 2 showing DLT.

If, unexpectedly, at least 2 patients are observed to have DLT at the initial dose level 0, then the next dose level evaluated will be the lowest dose level, -2, and further dose escalations to dose level -1 will proceed as outlined above from that dose level. If there is no RPTD declared, there will be no expansion to the phase II portion of the study. The phase I portion of the study will include between 9 and 12 patients depending upon the number of dose levels evaluated.

Phase II Study Design Phase II will follow a Simon's Optimal two-stage design to indicate proof of concept regarding the PFS rate of ixazomib in combination with ONC201 and Dexamethasone at the RPTD established in phase I. Once the RPTD for combination therapy has been established, an additional 24 patients will be enrolled for a total of 30 evaluable patients (24 + 6 from phase I at RPTD).

In considering a Simon's Optimal two-stage design, the plan is to look at each patient at 2 months after initiating study treatment (3 drug combination) and classify each patient as responder or non-responder at the 2 month time point. A responder is a patient who has stable disease or better (not progressed) since initiating study treatment; a non-responder is someone whose disease has progressed according to IMWG criteria. The population of relapsed and refractory MM patients in this study will likely all have progressed on standard therapy; therefore the null hypothesis being tested is that the disease control rate at 2 months is 5%. As per IMWG criteria, if patients show progression after 1 cycle of triplet therapy, they will continue on therapy and a repeat assessment will be performed after cycle 2 in order to confirm progression of disease.

Stage 1:

* Enroll 9 patients including the 6 patients being evaluated from the phase I portion of the study
* Evaluate patients at 2 months post initiation of treatment
* If 0 have responded (progression-free), i.e. if all 9 have progressed, then stop trial for futility and conclude that the proportion who will be progression-free at 2 months is less than 5%.
* If 1 or more have responded (progression-free) at 2 months, then proceed to Stage 2.

Stage 2:

* Enroll an additional 21 patients
* Evaluate patients at 2 months post initiation of treatment If 4 or more of the 30 patients have responded (progression-free) at 2 months then the null hypothesis is rejected and further investigation of this treatment combination is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent: Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care
* Target Population

  1. Symptomatic MM having progressed on 2 prior therapies including proteasome inhibitor (i.e. bortezomib, carfilzomib ixazomib), immunomodulatory drug (i.e., thalidomide, lenalidomide, pomalidomide), and daratumumab or other CD38 targeting monoclonal antibody. Proteasome inhibitor refractory patients are eligible. Subjects must not be candidates for treatment regimens known to provide clinical benefit to be eligible for this study.
  2. Male or female patients 18 years or older
  3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
  4. Patients must have measurable disease defined by at least 1 of the following 3 measurements:

  i. Serum M-protein > 0.5 g/dL ii. Urine M-protein > 200 mg/24 hours iii. Serum free light chain assay: involved free light chain level >10 mg/dL (> 100 mg/L) provided the serum free light chain ratio is abnormal

Exclusion Criteria:

* Medical History and Concurrent Diseases

  1. Peripheral neuropathy > Grade 2 or >Grade 1 with pain on clinical examination during the Screening period.
  2. Significant cardiac disease as determined by the investigator including:

  i. Known or suspected cardiac amyloidosis ii. Congestive heart failure of Class III or IV of the NYHA classification iii. Uncontrolled angina, hypertension or arrhythmia iv. Myocardial infarction in the past 6 months v. Any uncontrolled or severe cardiovascular disease vi. QTc > 470 milliseconds (msec) on a 12-lead ECG obtained during the Screening period. If a machine reading is above this value, the ECG should be reviewed by a qualified reader and confirmed on a subsequent ECG.

  c. Known active hepatitis B (defined as most recent serum PCR or hepatitis B surface antigen positive) or active hepatitis C (note, hepatitis C in sustained virologic response defined as negative RNA PCR at least 12 weeks after any therapy is permitted).

  d. Any medical conditions that, in the investigator's opinion, would impose excessive risk to the subject, e.g., any uncontrolled disease, such as pulmonary disease, infection, seizure disorder, uncontrolled hyperglycemia.

  e. Any altered mental status or any psychiatric condition that would interfere with the understanding of the informed consent or limit compliance with study requirements.

  f. Prior or concurrent malignancy, except for the following: i. Adequately treated basal cell or squamous cell skin cancer ii. Cervical carcinoma in situ iii. Adequately treated Stage I or II cancer from which the subject is currently in complete remission.

iv. Or any other cancer from which the subject has been disease-free for ≥ 3 years g. Diarrhea > Grade 1, based on the NCI CTCAE grading, in the absence of antidiarrheals.

h. Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of study drug, including difficulty swallowing.

i. Males or females of childbearing potential who do not agree to practice 2 effective methods of contraception, at the same time through 90 days after the last dose of study drug j. Females who are pregnant or breastfeeding. k. Diagnosis of Waldenstrom's macroglobulinemia, POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes) syndrome, plasma cell leukemia, myeloproliferative syndrome, or primary amyloidosis (with the exception of patients whose amyloidosis has been documented as a complication of MM, who will be evaluated on a case-by-case basis for trial participation).

l. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study drug administration.

m. Parkinson's disease 4) Physical and Laboratory Test Findings

a. Corrected serum calcium ≥ 14 mg/dl within 2 weeks of enrollment (despite appropriate measure such a short course of steroids, bisphosphonates, hydration, and calcitonin).

b. Absolute neutrophil count < 1000 cells/mm3. No growth factors allowed within 1 week of enrollment.

c. Platelets < 75,000 cell/mm3 (75 x 109/L). Qualifying laboratory value must occur at most recent measurement before enrollment and must be no more than 14 days before enrollment. No transfusions are allowed within 72 hours prior to study drug administration.

d. Hemoglobin < 8 g/dL. Qualifying laboratory value must occur at most recent measurement before enrollment and must be no more than 14 days before enrollment. No transfusions are allowed within 72 hours before qualifying laboratory value e. Serum bilirubin ≥ 1.5 x ULN, patients with Gilbert's syndrome and a total bilirubin of < 3 times ULN are permitted) f. AST or ALT ≥ 3 x ULN. g. CrCl < 30 ml/min/1.73m2. Creatinine clearance is estimated by the CKD-EPI formula. (Calculator available at https://www.kidney.org/professionals/kdoqi/gfr_calculator.)

* Prior Therapy or Surgery

  1. Major surgery or radiation therapy within 14 days before study drug administration.
  2. Kyphoplasty or vertebroplasty within 1 week of enrollment.
  3. Administration of chemotherapy, biological, immunotherapy, or investigational agent (therapeutic or diagnostic) within 3 weeks before enrollment (14 days for non-myelosuppressive therapy). Subjects should be 6 weeks from last dose of nitrosourea, nitrogen mustards or monoclonal antibody, 12 weeks from autologous SCT, and 16 weeks from allogeneic SCT.
  4. Corticosteroids use exceeding a cumulative dose of 160 mg of dexamethasone during screening.
  5. If prior allogeneic stem cell transplant, history of moderate to severe chronic graft versus host disease (GVHD).
  6. Treatment with plasmapheresis within 4 weeks before enrollment.
  7. NSAIDs, IV contrast, aminoglycosides, or other potentially nephrotoxic drugs within 2 weeks of enrollment.
  8. Current use of a non-standard dialysis membrane.
  9. Systemic treatment with strong inhibitors or inducers of CYP450 system should not be used on study including but not limited to fluvoxamine, enoxacin, ciprofloxacin, clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole, rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital, buproprion, fluoxetine, paroxetine, ticlopidine, or St. John's wort within 14 days before the first dose of study treatment. Ixazomib has significant drug-drug interactions with strong CYP3A inducers. No drug-drug interactions with the CYP450 screen have been found with ONC201, but the analysis of these studies is not complete, so during the study use of inhibitors or inducers of CYP450 system is excluded.
  10. Failure to have fully recovered (i.e., Grade 1 toxicity or less, with the exception of alopecia) from clinically significant effects of prior chemotherapy regardless of interval since last treatment.
* Allergies and Adverse Drug Reaction Known hypersensitivity to bortezomib, ixazomib, dexamethasone, ONC201

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose (RPTD) | 9 Months
  of triplet therapy (ixazomib + ONC201+ dexamethasone) following a 3+3 escalation design

SECONDARY OUTCOMES:
Disease control rate | 2 months
  2 month disease control rate defined as the proportion of patients that have stable or better disease after two months of treatment initiation according to IMWG criteria: Stable disease, partial remission, or complete remission
Progression free survival (PFS) | 6 months
  Median Progression free survival for the phase I and II patients treated at the recommended phase II dose. PFS is defined as the duration of time from start of treatment to the first occurrence of disease progression or death on study from any cause, whichever occurs earlier.
Duration of response (DOR) | 6 months
  Median duration of response for the phase I and II patients treated at the recommended phase II dose. DOR is defined as the time from first evidence of PR or better to confirmation of disease progression.
Clinical benefit rate (CBR) | 6 months
  Clinical benefit rate for the phase I and II patients treated at the recommended phase II dose level. CBR is the combination of the ORR and minimal response (MR) i.e. this includes sCR, CR, VGPR, PR, and MR.

CONTACTS AND LOCATIONS:
Overall Officials: Ajai Chari, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data and safety will be monitored using an internal Data and Safety Monitoring Plan (DSMP) led by the PI. Other members involved with the review will include sub-Investigators, the myeloma research program manager, and clinical research coordinators. All of these individuals have experience in the routine clinical care as well clinical research and monitoring of subjects with multiple myeloma. A statistician will also be involved with the review.